CLINICAL TRIAL: NCT02715960
Title: Pharmacogenomics Study on Treatment of Psoriasis Vulgaris by Acitretin Capsules
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Yijing He, Associate Professor, Central South University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016 AW/CSU/PS
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2015-12

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — Acitretin; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single-arm (Experimental): intervention: open registry, non-randomized, single-arm trial. Acitretin Capsules: 2.5 per piece.
  Interventions: Drug: Acitretin Capsules

INTERVENTIONS:
Drug: Acitretin Capsules — During The first treatment stage:10mg per day, 3 days,oral; The second stage: 20mg per day, 3 days,oral; The third stage: 30mg per day, and maintain this dose,oral.
  Other Names: Tretinoin, Vitamine A Acid

SUMMARY:
In an early clinical research, 138 patients completed the treatment of Psoriasis Vulgaris by Acitretin Capsules in 8 weeks, the results indicate 75 cases effectively (54.3%), 50 cases invalid(36.2%), 13 cases serious(9.4%). To investigate the influence of genetic factors on the curative effect and find the relationships between genetic variants and the response of Acitretin Capsules to treatment of Psoriasis Vulgaris.

DETAILED DESCRIPTION:
Investigators analyzed the various levels of genetic factors, including: 1.To analysis the key gene variants which associated with ADME affect the efficacy of Acitretin Capsules; 2.Direct full genetic sequencing of MHC genes, to explore the genetic variations of efficacy and side effects; 3. Direct sequencing of all exons in the gene in the patients of the response of serious and effectively, to explores the rare genetic variation may cause deterioration of treatment by Acitretin Capsules.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed according to Classification criteria for Psoriasis vulgaris
2. Patients aged 18 to 70 years (to the date of screening)
3. PASI grade ≥7point
4. Not treatment in the Topical corticosteroids, Immunosuppression, Biologicals agents or Tretinoin cream, Phototherapy nearly one months before enrolled.
5. Total bilirubin < 1.5 x ULN, AST(SGOT)/ALT(SGPT) <2.5 x ULN if not liver metastases<5 x ULN if known liver metastases, Creatinine clearance <1.5 x ULN
6. Understanding the whole process of the study, voluntary participation and signed the informed consent

Exclusion Criteria:

1. Pregnant women, ready to pregnant or lactating women
2. Have a serious heart, lung, kidney and other vital organs and endocrine system lesions and the history
3. Patients is liver function abnormal persons (ALT above the center laboratory normal limit) or hepatitis b patient grain carriers
4. Patients with chronic diarrhea, or peptic ulcer nearly 1 year
5. Patients suffering from malignant tumor
6. Patients suffering from acute and chronic infectious diseases
7. Mental disorders, history of alcohol abuse, drug or other substance abuse
8. Other cases which researchers believe that can not enroll

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
disease control rate | 8 weeks after the first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Chen, MD, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided
data not entered